CLINICAL TRIAL: NCT00684853
Title: Intravitreal Bevacizumab Combined With PDT (Full Fluence) Versus Bevacizumab to Treat Exudative Age-Related Macular Degeneration
Brief Title: Intravitreal Bevacizumab Combined With PDT Versus Bevacizumab to Treat Exudative AMD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Anderson Teixeira, MD, UNIFESP
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pep1
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Macular Degeneration
Keywords: AMD; PDT; Avastin; Bevacizumab; Full fluence; exudative; CNV; Drusen; ARMD; Vetaporfin; efficacy; treatment
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: bevacizumab; Drug: vetaporfin
- 2 (Active Comparator)
  Interventions: Drug: vetaporfin

INTERVENTIONS:
Drug: bevacizumab — 1.25 mg of bevacizumab intravitreal
  Arms: 1
Drug: vetaporfin — full fluence of vetaporfin

SUMMARY:
The purpose of this study is to determine the association of bevacizumab and PDT is safety and effective in the treatment of exudative AMD

DETAILED DESCRIPTION:
Exudative AMD is the leader of blind in people more than 60 years. The best treatment for this disease today are monthly injections of anti-VEGF in the vitreous cavity which increase the chance to get endophthalmites.

The participants of this study will be randomized in 1:1 ration to one of the two study groups: single therapy of bevacizumab (3 injections in 3 months) or association of bevacizumab (3 injections in 3 months) and full fluence of PDT (single at the baseline). All bevacizumab injection will contain 1.25g of the drug and will be administrate every month for 3 continuos months.

After randomization, participants will return to the clinic approximately every four weeks for 4 months for study assessments and possible re-treatment (if is necessary). Participants will return to the clinic at week 20 for a final study assessment. Study assessments include: visual acuity, optical coherence tomography and fundus photography.

ELIGIBILITY:
Inclusion Criteria:

* more or iqual 50 years old
* male or female
* Choroidal neovascularization sub or just foveal the fovea secondary to AMD (Predominantly Classic, Minimally Classic, and Occult lesions acceptable)
* Greatest linear dimension (GLD) of entire lesion < 5400 µm (no reading center confirmation required)
* ETDRS best corrected visual acuity of 20/40 - 20/320 (73 - 24 letter score)
* Total area of lesion must < 9 MPS DA

Exclusion Criteria:

* pre-treatment
* ETDRS best corrected visual acuity better than 34 letters
* macular surgery history
* laser photocoagulation in the study eye within 30 dais
* eye surgery within 30 days
* history of no-treat glaucoma
* acuite uveits
* history of endophthalmites
* vitreous hemorrhage
* geographic atrophy or fibrosis corresponding > 50% of the lesion

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The mean change in best-corrected ETDRS visual acuity in the study eye from baseline to 4 months | 4

SECONDARY OUTCOMES:
The overall probability of re-injection | 4
Proportion of participants with reduction in retinal thickening in the center subfield (i.e., thickness > 200 microns) of ³50% and of at least 50 microns from baseline | 4
Mean change in area of leakage, CNV and lesion by the FA and ICG | 4

CONTACTS AND LOCATIONS:
Locations (1):
- UNIFESP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Smith BT, Dhalla MS, Shah GK, Blinder KJ, Ryan EH Jr, Mittra RA. Intravitreal injection of bevacizumab combined with verteporfin photodynamic therapy for choroidal neovascularization in age-related macular degeneration. Retina. 2008 May;28(5):675-81. doi: 10.1097/IAE.0b013e31816b316e. PMID 18463509
- [Background] Colquitt JL, Jones J, Tan SC, Takeda A, Clegg AJ, Price A. Ranibizumab and pegaptanib for the treatment of age-related macular degeneration: a systematic review and economic evaluation. Health Technol Assess. 2008 May;12(16):iii-iv, ix-201. doi: 10.3310/hta12160. PMID 18462575
- [Background] Ahmadieh H, Taei R, Soheilian M, Riazi-Esfahani M, Ahadi H. Single-session photodynamic therapy combined with intravitreal bevacizumab for neovascular age-related macular degeneration. Eur J Ophthalmol. 2008 Mar-Apr;18(2):297-300. doi: 10.1177/112067210801800222. PMID 18320527
- [Background] Weigert G, Michels S, Sacu S, Varga A, Prager F, Geitzenauer W, Schmidt-Erfurth U. Intravitreal bevacizumab (Avastin) therapy versus photodynamic therapy plus intravitreal triamcinolone for neovascular age-related macular degeneration: 6-month results of a prospective, randomised, controlled clinical study. Br J Ophthalmol. 2008 Mar;92(3):356-60. doi: 10.1136/bjo.2007.125823. PMID 18303156
- [Background] Bashshur ZF, Schakal A, Hamam RN, El Haibi CP, Jaafar RF, Noureddin BN. Intravitreal bevacizumab vs verteporfin photodynamic therapy for neovascular age-related macular degeneration. Arch Ophthalmol. 2007 Oct;125(10):1357-61. doi: 10.1001/archopht.125.10.1357. PMID 17923543
- [Background] Ladas ID, Kotsolis AI, Papakostas TD, Rouvas AA, Karagiannis DA, Vergados I. Intravitreal bevacizumab combined with photodynamic therapy for the treatment of occult choroidal neovascularization associated with serous pigment epithelium detachment in age-related macular degeneration. Retina. 2007 Sep;27(7):891-6. doi: 10.1097/IAE.0b013e3180ca9ad9. PMID 17891013
- [Background] Ladewig MS, Karl SE, Hamelmann V, Helb HM, Scholl HP, Holz FG, Eter N. Combined intravitreal bevacizumab and photodynamic therapy for neovascular age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2008 Jan;246(1):17-25. doi: 10.1007/s00417-007-0654-x. Epub 2007 Aug 15. PMID 17701197
- [Background] Hahn R, Sacu S, Michels S, Varga A, Weigert G, Geitzenauer W, Vecsei-Marlovits P, Schmidt-Erfurth U. [Intravitreal bevacizumab versus verteporfin and intravitreal triamcinolone acetonide in patients with neovascular age-related macula degeneration]. Ophthalmologe. 2007 Jul;104(7):588-93. doi: 10.1007/s00347-007-1547-4. German. PMID 17564719
- [Background] Lazic R, Gabric N. Verteporfin therapy and intravitreal bevacizumab combined and alone in choroidal neovascularization due to age-related macular degeneration. Ophthalmology. 2007 Jun;114(6):1179-85. doi: 10.1016/j.ophtha.2007.03.006. PMID 17544776
- [Background] Lazic R, Gabric N, Dekaris I, Gavric M, Bosnar D. Photodynamic therapy combined with intravitreal bevacizumab (Avastin) in treatment of choroidal neovascularization secondary to age-related macular degeneration. Coll Antropol. 2007 Jan;31 Suppl 1:71-5. PMID 17469756
- [Background] Costa RA, Jorge R, Calucci D, Melo LA Jr, Cardillo JA, Scott IU. Intravitreal bevacizumab (Avastin) in combination with verteporfin photodynamic therapy for choroidal neovascularization associated with age-related macular degeneration (IBeVe Study). Graefes Arch Clin Exp Ophthalmol. 2007 Sep;245(9):1273-80. doi: 10.1007/s00417-007-0557-x. Epub 2007 Feb 28. PMID 17333238
- [Background] Augustin AJ, Puls S, Offermann I. Triple therapy for choroidal neovascularization due to age-related macular degeneration: verteporfin PDT, bevacizumab, and dexamethasone. Retina. 2007 Feb;27(2):133-40. doi: 10.1097/IAE.0b013e3180323de7. PMID 17290193